CLINICAL TRIAL: NCT01300078
Title: A Phase 1 Open Label, Randomized Clinical Trial Assessing Safety of MF101 for Hot Flushes and Menopausal Symptoms in Postmenopausal Women
Brief Title: A Clinical Trial Assessing Safety of MF101 for Hot Flushes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bionovo (Industry)
Responsible Party: Mary Tagliaferri, MD, LAc/President and CMO, Bionovo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF101-008
Record Dates: First submitted 2011-02-16; First posted 2011-02-21 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-06

CONDITIONS: Hot Flashes
Keywords: Hot Flashes; Hot Flushes; Vasomotor Symptoms; Menopausal Symptoms
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MF101 10 grams/day (Experimental)
  Interventions: Drug: MF101
- MF101 15 grams/day (Experimental)
  Interventions: Drug: MF101

INTERVENTIONS:
Drug: MF101 — MF101 10 g/day MF101 15 g/day
  Other Names: Menerba

SUMMARY:
This Phase 1, open label, randomized clinical trial will enroll 40 generally healthy, postmenopausal women aged 40-65 years old. Women will be randomized to one of two oral doses of MF101 for 4 weeks. Participants will be recruited at 3 clinical sites in the United States.

DETAILED DESCRIPTION:
MF101 is an oral, non-hormonal, botanical agent being investigated for the treatment of menopausal hot flashes.

ELIGIBILITY:
Inclusion Criteria (partial list):

* Postmenopausal women aged 40-65 years.
* Provide informed consent.
* Currently receive medical care from a health care provider. Other inclusions apply.

Exclusion Criteria (partial list):

* History of malignancy other than non-melanoma skin cancer or cervical cancer that was diagnosed and fully treated less than 5 years before screening.
* Unexplained uterine bleeding within 6 months prior to Screening.
* History of deep vein thrombosis or pulmonary embolism.
* Active liver disease or a history of impaired.
* Active gallbladder disease. Other exclusions apply.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of MF101, 10 g/day and 15 g/day | Randomization to 4 weeks
  New or worsening abnormalities on breast, physical and general exams, laboratory measures, transvaginal ultrasound, abnormal uterine bleeding, adverse events and serious adverse events.

SECONDARY OUTCOMES:
Compare the safety of MF101 10g/day and 15 g/day | Randomization to 4 Weeks
  To compare the safety of the 2 doses of MF101

CONTACTS AND LOCATIONS:
Overall Officials: Wulf Utian, PhD, DSc(Med), FRCOG, FACOG, Principal Investigator
Locations (4):
- United States (4):
  - Alta Bates, Jordan Research and Education Institute (REDI), Berkeley, California
  - Clinical Trials Research, Lincoln, California
  - Northern California Research, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California